CLINICAL TRIAL: NCT01556672
Title: Open-label Study on Small Bowel Lesions Suggestive of Crohn's Disease in Patients With Moderate to Severe Plaque Psoriasis Treated With Adalimumab
Brief Title: Adalimumab-psoriasis and Small Bowel Lesions
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Innovaderm Research Inc. (Other)
Collaborators: Abbott (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Inno-6021; IMM-11-0110 (Other Grant/Funding Number: Abbott)
Record Dates: First submitted 2012-03-15; First posted 2012-03-16 (Estimated); Last update posted 2016-06-29 (Estimated); Status verified 2016-06

CONDITIONS: Plaque Psoriasis; Crohn's Disease
Keywords: small bowel lesions; Crohn's Disease; Plaque psoriasis; adalimumab; capsule endoscopy
MeSH Terms: conditions — Crohn Disease | interventions — Adalimumab; Capsule Endoscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- adalimumab (Experimental): All patients will receive adalimumab 80 mg followed by 40 mg at week 1 and 40 mg every other week (EOW) thereafter.
  Interventions: Drug: Adalimumab; Device: Capsule endoscopy

INTERVENTIONS:
Drug: Adalimumab — Adalimumab will be administered sub-cutaneously to all patients entering the study with a loading dose of 80 mg followed by 40 mg at week 1 and 40 mg every other week. Patients who did not have small bowel lesions detected will be in the study and receive adalimumab until week 12. Patients who had small bowel lesions detected will be in the study and receive adalimumab until week 24.
  Other Names: Humira
Device: Capsule endoscopy — All patients will undergo capsule endoscopy (EndoCapsule EC type 1; Olympus) to treatment initiation (adalimumab) in order to detect the presence of small bowel lesions suggestive of Crohn's disease. Twenty-four (24) weeks after treatment with adalimumab was initiated, patients for whom small bowel lesions were detected will undergo a second capsule endoscopy to evaluate changes in bowel inflammation.
  Other Names: EndoCapsule EC-1; OLYMPUS EC TYPE 1

SUMMARY:
This study will determine the prevalence of small bowel lesions suggestive of Crohn's disease (CD) in patients with moderate to severe plaque psoriasis using capsule endoscopy. The study also aims to determine if the treatment of psoriasis with adalimumab will have an effect on the healing of the small bowel for patients who have lesions suggestive of CD.

Patients with psoriasis are at increased risk of developing Crohn's disease (CD), but the exact prevalence of CD in patients with psoriasis at this time is unknown as many patients probably have undiagnosed disease as the early signs will often cause no symptoms. CD is therefore receiving very little attention from dermatologists who are treating patients with psoriasis. For example, very few dermatologists will actively question patients with psoriasis about symptoms of CD. This lack of knowledge may induce delays in diagnosis. By the time the diagnosis is made and patients receive their first treatment, they may already have significant fibrosis and stenosis of the intestine. Current treatments, including adalimumab, cannot reverse small bowel anomalies to normal in the presence of fibrosis. Therefore, many patients with a late diagnosis will still have symptoms or will eventually require surgery despite good control of the inflammation. Treatment of CD should start as early as possible, as early treatment has been associated with an increased rate of complete healing. Complete control of the disease at its early stages may prevent complications.

DETAILED DESCRIPTION:
This open-label, phase IV, 24-week study will recruit a total of 100 patients with moderate to severe plaque psoriasis without a diagnosis of inflammatory bowel disease. All patients will undergo capsule endoscopy at the beginning of the study to detect the presence of small bowel lesions suggestive of CD such as erosions and ulcers. All patients will receive adalimumab 80 mg followed by 40 mg at week 1 and 40 mg every other week (EOW) thereafter. Patients for whom no small bowel lesions suggestive of CD were detected will remain in the study and under adalimumab therapy until week 12. A second capsule endoscopy will be performed 24 weeks after initiation of adalimumab for patients who had small bowel lesions suggestive of CD to evaluate changes in bowel inflammation.

ELIGIBILITY:
Inclusion Criteria:

* Men or women are 18 to 80 years of age at time of consent
* At least a 6-month history of chronic moderate to severe plaque psoriasis and is a candidate for systemic therapy
* BSA covered with psoriasis of at least 5% or more at Day 0
* Unless subject or subject's partner is in a menopausal state for at least a year, surgically sterile, clinically diagnosed infertile, having a same-sex partner or abstinent, female of childbearing potential or male patient (or his partner) is willing to use effective contraceptive method for at least 30 days before Day 0 and at least 6 months after the last study drug administration
* Is judged not to have contraindications to adalimumab as determined by the principal investigator based upon the results of medical history, laboratory profile, physical examination and chest X ray (CXR) performed at screening
* Negative results for latent TB infection with a PPD or QuantiFERON®-TB Gold test and a CXR
* Capable of giving informed consent and the consent must be obtained prior to any study related procedures
* Must be able and willing to self-administer SC injections or have a qualified person available to administer SC injections

Exclusion Criteria:

* Diagnosis of inflammatory bowel's disease
* Presence of any evidence of gastrointestinal obstruction, strictures and/or fistulas
* Presence of highly suspected or documented gastroparesis
* Known presence of gastrointestinal motility disorders
* Known presence of delayed gastric emptying
* Prior abdominal surgery of the gastrointestinal tract other than uncomplicated procedures that would be unlikely to lead to bowel obstruction based on the clinical judgment of the investigator
* Presence of pacemaker, defibrillator or other electromedical device
* Expected to undergo a MRI examination within 7 days after ingestion of the capsule
* Swallowing disorder
* Presence of other skin diseases or skin infections that may interfere with evaluation of psoriasis or with patient's safety at Day 0
* History of an allergic reaction or significant sensitivity to constituents of study drug, including latex
* Use of any biological therapy for the treatment of psoriasis less than 90 days before Day 0
* Use of any other non-biological systemic therapy for the treatment of psoriasis within 28 days before Day 0
* Is planning to intentionally increase exposure to ultraviolet light at any time during the study period
* Is taking or requires systemic (i.e., oral or injectable) corticosteroids within 28 days of Day 0 or during the study
* Used any topical treatments for psoriasis or phototherapy within two weeks prior to Day 0
* Received Anakinra/Kineret within the last 2 weeks prior to Day 0
* Used any investigational non-biological agent within 30 days prior to Day 0, or within 5 half lives of the investigational agent prior to day 0
* Used NSAIDs for 28 days before Day 0
* Has a poorly controlled medical condition in the opinion of the investigator, would put the patient at risk if participating in the study
* Multiple sclerosis or presents with or has a history of neurologic symptoms suggestive of CNS demyelinating disease
* Current signs or symptoms of or a history of systemic lupus erythematosus or lupus like syndrome
* History of cancer or lymphoproliferative disease other than a successfully treated non metastatic cutaneous squamous cell or basal cell carcinoma and/or localized carcinoma in situ of the cervix
* History of listeriosis, treated or untreated TB, persistent chronic infections, or recent active infections requiring hospitalization or treatment with intravenous anti-infectives within 30 days or oral anti-infectives within 14 days prior to Day 0
* Received any live attenuated vaccine 28 days or less before Day 0 or plans to receive one during the study
* Hepatitis B or hepatitis C
* Clinically significant abnormal results for hemoglobin, white blood cell count, platelet count, ALT, AST, total bilirubin or creatinine
* Current use or plan to use anti-retroviral therapy at any time during the study
* Known immune deficiency or is immunocompromised
* Current pregnancy or lactation or considering becoming pregnant during the study or for 150 days after the last dose of study medication
* History of clinically significant drug or alcohol abuse in the last year
* Is considered by the investigator, for any reason, to be an unsuitable candidate for the study

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2012-04; Primary Completion 2016-01 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Prevalence of small bowel lesions suggestive of Crohn's disease in patients with moderate to severe plaque psoriasis as visualized by capsule endoscopy | Day 0

SECONDARY OUTCOMES:
Induction of mucosal healing at week 24 after initiation of adalimumab in patients with small bowel lesions suggestive of Crohn's disease and psoriasis as defined by absence of villous edema, erosions and ulcers | 24 weeks
Study the relationship between mucosal healing and plaque psoriasis improvement in patients with small bowel lesions suggestive of Crohn's disease and psoriasis | 24 weeks
  as evaluated by the absence of villous edema, erosions and ulcers and mean change from baseline in PASI at week 24
Study the relationship between levels of fecal calprotectin and endoscopy findings | Day 0 and week 24
Change from baseline in PASI at Week 12 for patients who had presence of small bowel lesions suggestive of CD as compared to patients who did not have small bowel lesions suggestive of CD | 12 weeks
Proportion of patients reaching Psoriasis Area and Severity Index (PASI) 75 at Week 12 for patients who had small bowel lesions suggestive of CD as compared to patients who did not have small bowel lesions suggestive of CD. | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Robert Bissonnette, MD, FRCPC, Principal Investigator — Innovaderm Research Inc.
Locations (3):
- Canada (3):
  - Lynderm Research, Markham, Ontario
  - Innovaderm Research Inc., Montreal, Quebec
  - Dr Isabelle Delorme, Saint-Hyacinthe, Quebec

IPD SHARING:
Plan to Share IPD: No